CLINICAL TRIAL: NCT04118049
Title: The Effect of Vaginal Probiotics on the Vaginal Microenvironment in Patients Using Vaginal Pessaries: a Randomized Controlled Trial.
Brief Title: Vaginal Probiotics and Pessaries and Their Impact on the Vaginal Microenvironment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: University of Maryland (Other); University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R-HHC-2019-0069
Record Dates: First submitted 2019-10-01; First posted 2019-10-07 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Pelvic Organ Prolapse; Inflammatory Response; Dysbiosis
Keywords: Pessary use; Probiotics; Cytokines; Microenvironment
MeSH Terms: conditions — Pelvic Organ Prolapse; Dysbiosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the treatment arm versus standard care arm.
Who Masked: Outcomes Assessor
Masking Description: Investigators performing vaginal specimens are blinded to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Probiotic Arm (Experimental): BiopHreshTM vaginal probiotic supplement (Good Clean Love, Inc. Eugene, OR) is offered over the counter. It contains a total of 5 billion lactobacilli: L. crispatus, L. gasseri, L. jensenii, and L. rhamnosus.
  RestoreTM gel: moisturizing personal lubricant.
  We will recommend to participants to use the probiotic supplement and vaginal lubricant as a vaginal suppository three times weekly at night for 3 months.
  Interventions: Other: BiopHreshTM vaginal probiotic supplement (Good Clean Love, Inc. Eugene, OR) and RestoreTM gel.
- Standard Care Arm (Other): Women will perform standard care which includes follow up at 3 months for pessary removal/care.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: BiopHreshTM vaginal probiotic supplement (Good Clean Love, Inc. Eugene, OR) and RestoreTM gel. — BiopHreshTM is a vaginal probiotic supplement that is offered over the counter and contains four different lactobacilli strains (L. crispatus, L. gasseri, L. jensenii, and L. rhamnosus). RestoreTM is a moisturizing personal lubricant that has been on the market for three years. Participants will use 1 probiotic capsule with RestoreTM gel nightly three times weekly.
  Arms: Vaginal Probiotic Arm
Other: Standard Care — Standard care arm is standard care for pessary use. Pessary maintenance will be performed standardly by their provider.
  Arms: Standard Care Arm

SUMMARY:
In this study, the investigators are evaluating the effect of vaginal probiotics on the bothersome side effects of pessary use and the impact on the vaginal microenvironment (lactobacilli, anaerobic bacteria, mobiluncus bacteria, WBCs, cellular debris, epithelial cells, and BVAB-1), and inflammatory environment (cytokines).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (no menstruation >12 months)
* Subjects presenting for 2 week post initial pessary insertion appointment or presenting for routine pessary care follow up appointment
* Planning on continuing to use a pessary for treatment for at least 3 months
* Pessary maintenance performed by provider (as opposed to self-care)
* Able to understand English
* Able/willing to sign informed consent document

Exclusion Criteria:

* Lack of cognitive ability to consent to participate in study and to complete the questionnaires
* Planned prolapse surgery less than 3 months from enrollment
* Presence of vaginal fistulas
* Pessary self-care (patient changes and cleans her own pessary)
* Receiving immunosuppressive therapy or history of immunodeficiency
* Presence of an indwelling vascular access line or structural heart disease
* Within 6 weeks from any abdominal or pelvic surgery or other major surgery
* Allergy to lactobacillus (contents of probiotic)
* Allergy to beta-lactam antibiotics, erythromycin and clindamycin
* Use of any probiotic pills, creams, or suppositories currently

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change in vaginal microenvironment | Vaginal specimen assessment with gram stain will be assessed upon enrollment and after 3 months of treatment.
  Change in vaginal microenvironment on gram stain measuring lactobacilli, anaerobic bacteria, and mobiluncus, WBCs and epithelial cell maturation reported as Nugent Subscore.

SECONDARY OUTCOMES:
Pelvic Floor Disability Index (PFDI-20) | Participants will complete the PFDI-20 upon enrollment and after 3 months of treatment.
  The PFDI-20 will be used in order to evaluate pelvic floor symptoms.
Vaginal probiotic feasibility, compliance with, and side effects of probiotic use. | Participants will complete after 1 month of use as well as at 3 months.
  Unvalidated questionnaires (vaginal products and hromonal therapy questionnaire, subjective vaginal experiences over the past month questionnaire, and a vaginal probiotic questionnaire) were created in order to evaluate participant experiences with vaginal probiotics including feasibility, impact on symptoms from pessary use, and side effects from use. These questionnaires do not have scales.
Urinary tract infection incidence | During participant involvement in the study 3-4 months.
  Occurrences of urinary tract infections during the study period will be monitored.
BVAB-1 | Vaginal specimen will collect from participants upon enrollment and after 3 months.
  Evaluate the incidence of BVAB-1 and impact of vaginal probiotics on BVAB-1 in postmenopausal women via gram stain.
Pro-inflammatory cytokines (Interleukin (IL-6)), Tumor Necrosis Factor-alpha (TNF-alpha), Interleukin(IL-1alpha) and Interleukin (IL-1beta) | Vaginal specimens will be collected for cytokine analysis at enrollment and after 3 months
  Pro-inflammatory cytokines will be evaluated from vaginal specimens collected in order to evaluate (1) the impact of probiotics on the inflammatory environment of the vagina (2) longitudinal assessment of pro-inflammatory cytokines in pessary wearing patients.
Incidence of adverse events (safety and tolerability) | from enrollment to 3 month follow up visit
  number of adverse events (vaginal irritation)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Sappenfield, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sappenfield EC, Mellen C, Wilcox J, O'Hanlon DE, O'Sullivan DM, Tunitsky-Bitton E. The Impact of Vaginal Probiotics on Pessary Use: A Randomized Controlled Trial. Urogynecology (Phila). 2024 Jan 1;30(1):50-58. doi: 10.1097/SPV.0000000000001379. Epub 2023 Jul 18. PMID 37493229